CLINICAL TRIAL: NCT06795035
Title: ConMicro STEMI: Assessment of Coronary Microvascular Dysfunction After ST-Elevation Myocardial Infarction Using Continuous Saline Thermodilution
Brief Title: Assessment of Coronary Microvascular Dysfunction After STEMI Using Continuous Saline Thermodilution
Acronym: ConMICRO STEMI
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Khaled Ziada, MD, Interventional Cardiologist, The Cleveland Clinic
Other Study IDs: 25-015
Record Dates: First submitted 2025-01-24; First posted 2025-01-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: ST Elevation Myocardial Infarction; Coronary Microvascular Dysfunction; Microvascular Obstruction
Keywords: STEMI; Microvascular; MVO; MRR; Thermodilution
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Continuous Saline Thermodilution — Continuous saline thermodilution for determination of microvascular resistance reserve (MRR) is a novel operator-independent method to assess coronary microvascular function. CST has been studied in the setting of angina with nonobstructive coronary arteries (ANOCA), but not in the setting of acute MI. In contrast, bolus thermodilution, used to determine the index of microcirculatory resistance (IMR), has been shown in the setting of STEMI to predict extent of myocardial injury and long-term clinical outcomes (e.g., heart failure, mortality, nonfatal MI, and ischemic stroke). In contrast to bolus thermodilution techniques, CST does not require the use of active medications (e.g., papaverine or adenosine) -- only a small volume of normal saline.

SUMMARY:
The goal of this observational study to measure the heart's microvascular function in the setting of a myocardial infarction (MI), or heart attack, using a method called continuous saline thermodilution (CST). The participants will include people who are experiencing MI from sudden and complete blockage of a coronary artery requiring immediate balloon and/or stent therapy. After getting the balloon and/or stent therapy, participants will have their heart's microvascular system tested using CST. The main questions it aims to answer are:

* What measurements using CST can we expect from the heart's microvascular system during a treated MI?
* Can CST measurements during a treated MI predict the amount of heart muscle that is injured and that recovers?

For this study, participants will undergo measurement of their heart's microvascular function after balloon and/or stent therapy for the MI. They will then receive an MRI scan of the heart several days after the MI.

DETAILED DESCRIPTION:
This will be a non-interventional, prospective, descriptive analysis on a cohort of patients experiencing ST-elevation myocardial infarction (STEMI) who present to the Cleveland Clinic cardiac catheterization laboratory (CCL) for emergent primary percutaneous coronary intervention (PCI). The aim is to study acute coronary microvascular dysfunction using the method of continuous saline thermodilution to provide absolute measurements of coronary blood flow, coronary microvascular resistance, and microvascular resistance reserve (MRR) following primary PCI for STEMI patients.

Adult patients experiencing acute STEMI who present to the catheterization laboratory for emergent cardiac catheterization for STEMI, <24 hours after symptom onset, who undergo primary PCI to an IRA. Only those able to provide initial oral consent upon CCL presentation and confirmatory written consent following cardiac catheterization will be included in the study.

Study endpoints are part of usual standard practice, and include clinic visits with updated medical histories and physical examination, and echocardiography. Clinical endpoints of interest will include mortality, incident heart failure, anginal symptoms, and standard major adverse cardiac events including cardiac death, nonfatal MI, urgent coronary revascularization, or hospitalization for unstable angina.

ELIGIBILITY:
Inclusion Criteria:

* Adults (persons >18 years old) presenting to Cleveland Clinic cardiac catheterization lab within 24 hours of symptom onset, with clinical and EKG findings concerning for STEMI, with intent to undergo emergent primary PCI, who have culprit artery identified on diagnostic angiography
* Adults (persons >18 years old) presenting to Cleveland Clinic cardiac catheterization lab for pharmaco-invasive management of failed fibrinolysis, with intent to undergo emergent PCI, who have culprit artery identified on diagnostic angiography
* On-call treating interventional cardiologist is trained in the method of continuous saline thermodilution for coronary microvascular assessment

Exclusion Criteria:

* No evidence of coronary obstruction on diagnostic angiography (e.g., Takotsubo, myocarditis leading to STEMI activation).
* Patients in hemodynamic shock
* Culprit artery <3.0 mm in diameter.
* Culprit artery being a bypass graft
* Patients physically unable to tolerate additional time required to conduct coronary microvascular testing after primary PCI.
* Patients with eGFR <30 mL/min/1.73m2 are excluded from contributing cardiac MRI data
* Patients with standard contraindications to CMR (e.g., pacemakers, cochlear implants, certain prosthetic heart valves, certain surgical implants) are excluded from contributing cardiac MRI data
* Unable to provide verbal and written consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to catheterization lab within 24 hours of ischemic symptom onset with intent for emergent primary PCI due to STEMI on ECG or who have failed thrombolytic therapy and present for pharmaco-invasive management of STEMI.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Microvascular resistance reserve (MRR) | At enrollment
  Calculated index to assess coronary microvascular dysfunction (Q_hyperemia/Q_rest)*(Pa_rest/Pd_hyperemia)

SECONDARY OUTCOMES:
Change in LV Wall Motion Summed Score | From 1-day echo to 3-month routine follow up echo
  Global wall motion abnormality score by echo based on 16 segment model (0= normal, 1=mild hypokinetic, 2= hypokinetic, 3= severely hypokinetic, 4= akinetic, 5= aneurysmal)
Change in LVEF | From 1-day echo to 3-month routine follow up echo
  Left ventricular ejection fraction as quantified by routine baseline echo to routine follow up echo
Presence of microvascular obstruction | Within 3 days of hospital discharge
  Presence of microvascular obstruction on cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Ziada, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No